CLINICAL TRIAL: NCT01173835
Title: Incentive-based Intervention for Smoking Cessation and Prevention in High Schools
Acronym: Rise Above
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Suchitra Krishnan-Sarin, Associate Professor, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0902004736; R01DA026450 (NIH)
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: Tobacco Prevention and Cessation
Keywords: Adolescent tobacco use; Tobacco Free and Win; Incentive-based intervention; Contingency Management; Smoking Prevention; Smoking cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Forkhead Box Protein M1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Incentives for being tobacco free — Students who join the program will be entered into regularly scheduled drawings throughout the school year to earn incentives for being tobacco free.
  Other Names: Incentive-based program; Tobacco Free and Win; Contingency Management

SUMMARY:
The purpose of this study is to design an incentive-based intervention to motivate a tobacco-free lifestyle among high school students and to pilot the intervention in the first academic year in two schools (CT and NY) and examine feasibility and acceptability. Preliminary efficacy of the intervention will be assessed by implementing it in two new schools (CT and NY) in the second academic year and determine an effect size estimate for a larger trial.

The study is intended to assess the number of students joining the program and pledging to be smoke-free and to examine changes in tobacco use rates and attitudes following intervention exposure. We hypothesize that the schools will have lower rates of tobacco use and improvement in attitudes, norms and behavioral control over tobacco use after participating in the program.

ELIGIBILITY:
Inclusion Criteria:

* high school student at school that is invited to participate

Exclusion Criteria:

* no exclusion criteria

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1651 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The number of students who join the tobacco free program | at the end of each academic year

SECONDARY OUTCOMES:
Change in tobacco use rates and attitudes following the intervention exposure | at the end of each academic year

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, Ph.D., Principal Investigator — Yale University
Locations (1):
- CMHC, Substance Abuse Center, New Haven, Connecticut, United States